CLINICAL TRIAL: NCT06827886
Title: GPNMB-targeting Chimeric Antigen Receptor T-Cell Therapy (GCAR1) for a Patient With Alveolar Soft Part Sarcoma (CLIC-YYC-GPNMB-01)
Brief Title: GPNMB-targeting Chimeric Antigen Receptor T-Cell Therapy (GCAR1) for a Patient With Alveolar Soft Part Sarcoma
Acronym: GCAR1
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIC-YYC-GPNMB-01
Record Dates: First submitted 2025-02-03; First posted 2025-02-14 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Alveolar Soft Part Sarcoma
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part

STUDY DESIGN:
Intervention Model Description: Single Patient Study (SPS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GCAR1 (Experimental): GCAR1, a patient-specific cell therapy product containing a mixture of autologous lymphocytes transduced with a lentiviral vector containing a chimeric antigen receptor (CAR) that enables the specific targeting towards tumor cells expressing the cell surface protein glycoprotein non-metastatic B (GPNMB)
  Interventions: Biological: GCAR1

INTERVENTIONS:
Biological: GCAR1 — GCAR 1 is a patient-specific cell therapy product containing a mixture of autologous lymphocytes transduced with a lentiviral vector containing a chimeric antigen receptor (CAR) that enables the specific targeting towards tumor cells expressing the cell surface protein glycoprotein non-metastatic B (GPNMB).

SUMMARY:
CLIC-YYC-GPNMB-01 is a Single Patient Study (SPS) developed according to the Health Canada template and guidelines released in 2019 for studies to access therapies not otherwise available to patients, in the situation where there are no options of treatment or cure remaining. The patient under consideration for CLIC-YYC-GPNMB-01 has progressive metastatic alveolar soft part sarcoma (ASPS). The investigators propose to treat the patient with GCAR1, a patient-specific cell therapy product containing a mixture of autologous lymphocytes transduced with a lentiviral vector containing a chimeric antigen receptor (CAR) that enables the specific targeting towards tumor cells expressing the cell surface protein glycoprotein non-metastatic B (GPNMB).

ELIGIBILITY:
Inclusion Criteria:

1. Completion of Informed Consent Form

Exclusion Criteria:

1. Any significant medical issue(s) that would, in the opinion of the Principal Investigator (PI), prevent this patient from being dosed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Assess safety of GCAR1 | 1 year
  Treatment-Related Adverse Events to GCAR1 will be determined by monitoring participant for complications related to treatment using CTCAE v5.0.
Assess for anti-tumor activity | 1 year
  To assess for anti-tumor activity by measuring response of specified lesions. Response will be assessed by RECIST 1.1. Progression free survival (PFS) is calculated as the period from the day of starting administration of the study drug to the date that disease progression is confirmed by radiographic assessment. Diagnostic imaging (CT and/or MRI) will be performed pre-infusion to document measurable disease, and 4-6 weeks after GCAR1 T-cell infusion to evaluate response to therapy. If diagnostic imaging studies are performed at other times, either during or after treatment on this study, that data will be collected and information gained may be used to for further direction in the study of anti-GPNMB CAR T-cells, if appropriate consent is obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Shafey, MD, FRCPC, Principal Investigator — Alberta Health services
Locations (1):
- Tom Baker Cancer Centre/Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Canada

IPD SHARING:
Plan to Share IPD: No